CLINICAL TRIAL: NCT01947751
Title: Comparison Between Catheter Early Withdrawal or Maintenance in Sepsis or Septic Shock With Undefined Origin
Brief Title: Catheter Early Withdrawal or Maintenance in Sepsis or Septic Shock
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hospital Nossa Senhora da Conceicao (Other)
Responsible Party: Principal Investigator, Marcio Manozzo Boniatti, Principal investigator, Hospital Nossa Senhora da Conceicao
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HNSConceicao; HNSC022014 (Registry Identifier: 022014)
Record Dates: First submitted 2013-09-18; First posted 2013-09-20 (Estimated); Last update posted 2013-09-20 (Estimated); Status verified 2013-09

CONDITIONS: Catheter Related Infection
Keywords: Catheter related infection; Central venous catheter; CVC infection
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- CVC exchange (Active Comparator): The CVC will be removed immediately.
  Interventions: Procedure: CVC exchange
- CVC maintenance (Experimental): The CVC will be maintained, and exchanged only if confirmed catheter-related infection or worsening of sepsis
  Interventions: Drug: CVC maintenance

INTERVENTIONS:
Procedure: CVC exchange — CVC exchange when related infection is suspected
  Arms: CVC exchange
Drug: CVC maintenance — CVC maintenance and adding antibiotic therapy when related infection is suspected, waiting for the cultures to take the decision of changing CVC
  Other Names: Watchful waiting strategy
  Arms: CVC maintenance

SUMMARY:
Central venous catheter(CVC)-related infection is an inherent complication of this device that should be treated promptly. However, there are doubts about the need for the immediate withdrawal of CVC while there is still no confirmation of such infection. The aim of this study is to compare the resolution of CVC-related infection, testing two approaches: catheter´s early exchange, when the possibility of related sepsis is considered, versus the maintenance of the CVC and early antibiotic therapy until the infection is confirmed.

DETAILED DESCRIPTION:
The aim of this study is to compare the strategy of immediate removal of the catheter with a conservative strategy in resolution of infection in patients with sepsis or septic shock without a defined origin. The investigators intend to demonstrate that the conservative strategy can reduce the rate of unnecessary catheter removal, without increasing morbidity.

In the intervention group the investigators will adopt the conservative strategy, changing the CVC after the confirmation of infection related to it or non-improvement of sepsis. The control group is represented by the patients in whom the CVC is removed early.

ELIGIBILITY:
Inclusion Criteria:

* All patients with 18 years or more, admitted to ICU that had a CVC inserted before or after ICU admission and with infection with undefined origin.

Exclusion Criteria:

* Less than 18 years, severe neutropenia (<500/mm³), intravascular device (pacemaker, prosthetic valve), unequivocal signs of infection on the site of CVC insertion, patients who were terminally ill defined, bacteremia without a known source, refusal to signing the informed consent.

Ages: 18 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2013-03; Primary Completion 2014-01 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Infection resolution | 4 weeks
  Compare the resolution of CVC-related infection between the group that had the CVC exchanged, versus the CVC-maintenance plus adding antibiotics therapy group.

SECONDARY OUTCOMES:
Clinical variables | 6 months
  Comparison of PCR, leukocytes, temperature, length of stay and mortality in the two groups, as well as complication rates and number of catheters removed.

CONTACTS AND LOCATIONS:
Overall Officials: Marcio M Boniatti, PhD, Principal Investigator — Hospital Nossa Senhora da Conceicao
Locations (1):
- Hospital Nossa Senhora da Conceicao, Porto Alegre, Rio Grande do Sul, Brazil